CLINICAL TRIAL: NCT05328817
Title: Azithromycin Versus Erythromycin For Preterm Prelabor Rupture of Membranes: A Randomized Controlled Trial
Brief Title: Azithromycin Versus Erythromycin For Preterm Prelabor Rupture of Membranes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eastern Virginia Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-01-FB-0001
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Preterm Premature Rupture of Membrane
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Intervention Model Description: In order to maintain balanced groups, block randomization will be used. Pregnant women will be randomized in blocks of 6 with a total number of blocks to be 40. This will be conducted using STATA16 software, which will generate random permutations of sequential IDs of eligible study participants and their assignment to the treatment arms. This will be transferred to the REDCap in which a database will be created to facilitate random assignment during recruitment while maintaining concealment of randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erythromycin (Experimental): Receive 1) erythromycin 250 mg iv every 6 hours for 48 hours followed by 333 mg orally (pills) every 8 hours for 5 days
  Interventions: Drug: Antibiotics
- Azithromycin (Experimental): Receive azithromycin 500 mg iv daily for 48 hours followed by 500 mg orally (pills) for 5 days.
  Interventions: Drug: Antibiotics

INTERVENTIONS:
Drug: Antibiotics — In the absence of labor, broad-spectrum antibiotics (often called latency antibiotics) are recommended for women with PPROM less than 34 weeks to reduce chorioamnionitis, prolong latency, and decrease neonatal sepsis (12,13).
  Other Names: Latency antibiotics; Broad-spectrum antibiotics

SUMMARY:
Aim 1. To examine the latency period according to antibiotic regimens (erythromycin iv for two days followed by orally for 5 days vs. azithromycin iv for 2 days followed by 5 days orally).

Aim 2. To examine the latency period according to races stratified by antibiotic regimens.

Aim 3: To examine if there is a difference in neonatal morbidity and mortality stratified by antibiotic regimen.

DETAILED DESCRIPTION:
Significant differences exist in the pharmacokinetics and pharmacodynamics pathways of macrolide antibiotics between different races and ethnicities. Erythromycin compared to azithromycin interacts with more proteins and is likely affected by genetic variation. Therefore, the investigators hypothesize that the optimal latency antibiotic regimens for PPROM could potentially differ between races.

Due to the paucity of data regarding the use of an azithromycin regimen for latency antibiotics, the Eastern Virginia Medical School MFM team uses an erythromycin regimen even though azithromycin requires less frequent dosing, has lower rates of side effects, and is more cost effective. The Center for Maternal and Child Health Equity at Eastern Virginia Medical School was developed to address health disparities for mothers and their children, and the investigator team is committed to working with the center to address this research gap regarding latency antibiotic use in PPROM.

The aim is to determine the optimal antibiotic regimen for women with PPROM. The hypothesis to be tested are 1) The antibiotic regimen with azithromycin (iv for 2 days followed by 5 days orally) is associated with a longer latency period compared to the antibiotic regimen with erythromycin, and 2) The antibiotic regimen with azithromycin reduces disparity in latency period compared to the antibiotic regimen with erythromycin.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* PPROM from 22 weeks 0 days to 31 weeks 6 days at Sentara Norfolk General Hospital
* Membrane rupture within 36 hours of randomization, cervical dilation 3 cm or less, and 4 or fewer contractions in the 60-minutes monitoring before randomization

Exclusion Criteria:

* Non-reassuring fetal heart tracing
* Vaginal bleeding
* Indications for delivery
* Received any antibiotic therapy within 7 days other than initiation of Ampicillin treatment as part of latency antibiotics prior to transfer to Sentara Norfolk General Hospital
* Allergy to penicillin, erythromycin, or azithromycin

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Latency Period | At delivery
  The time interval between the first antibiotic dose to time of delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Tetsuya Kawakita, MD, Principal Investigator — Eastern Virginia Medical School

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Waters TP, Mercer B. Preterm PROM: prediction, prevention, principles. Clin Obstet Gynecol. 2011 Jun;54(2):307-12. doi: 10.1097/GRF.0b013e318217d4d3. PMID 21508700
- [Background] Meis PJ, Ernest JM, Moore ML. Causes of low birth weight births in public and private patients. Am J Obstet Gynecol. 1987 May;156(5):1165-8. doi: 10.1016/0002-9378(87)90133-5. PMID 3578431
- [Background] Beydoun SN, Yasin SY. Premature rupture of the membranes before 28 weeks: conservative management. Am J Obstet Gynecol. 1986 Sep;155(3):471-9. doi: 10.1016/0002-9378(86)90257-7. PMID 3752169
- [Background] Garite TJ, Freeman RK. Chorioamnionitis in the preterm gestation. Obstet Gynecol. 1982 May;59(5):539-45. PMID 7070724
- [Background] Pergialiotis V, Bellos I, Fanaki M, Antsaklis A, Loutradis D, Daskalakis G. The impact of residual oligohydramnios following preterm premature rupture of membranes on adverse pregnancy outcomes: a meta-analysis. Am J Obstet Gynecol. 2020 Jun;222(6):628-630. doi: 10.1016/j.ajog.2020.02.022. Epub 2020 Feb 25. No abstract available. PMID 32109463
- [Background] Costeloe KL, Hennessy EM, Haider S, Stacey F, Marlow N, Draper ES. Short term outcomes after extreme preterm birth in England: comparison of two birth cohorts in 1995 and 2006 (the EPICure studies). BMJ. 2012 Dec 4;345:e7976. doi: 10.1136/bmj.e7976. PMID 23212881
- [Background] Marlow N, Wolke D, Bracewell MA, Samara M; EPICure Study Group. Neurologic and developmental disability at six years of age after extremely preterm birth. N Engl J Med. 2005 Jan 6;352(1):9-19. doi: 10.1056/NEJMoa041367. PMID 15635108
- [Background] Averbuch B, Mazor M, Shoham-Vardi I, Chaim W, Vardi H, Horowitz S, Shuster M. Intra-uterine infection in women with preterm premature rupture of membranes: maternal and neonatal characteristics. Eur J Obstet Gynecol Reprod Biol. 1995 Sep;62(1):25-9. doi: 10.1016/0301-2115(95)02176-8. PMID 7493703
- [Background] Shen TT, DeFranco EA, Stamilio DM, Chang JJ, Muglia LJ. A population-based study of race-specific risk for preterm premature rupture of membranes. Am J Obstet Gynecol. 2008 Oct;199(4):373.e1-7. doi: 10.1016/j.ajog.2008.05.011. Epub 2008 Jul 29. PMID 18667175
- [Background] Drassinower D, Friedman AM, Obican SG, Levin H, Gyamfi-Bannerman C. Prolonged latency of preterm prelabour rupture of membranes and neurodevelopmental outcomes: a secondary analysis. BJOG. 2016 Sep;123(10):1629-35. doi: 10.1111/1471-0528.14133. Epub 2016 May 31. PMID 27245741
- [Background] Boghossian NS, Geraci M, Lorch SA, Phibbs CS, Edwards EM, Horbar JD. Racial and Ethnic Differences Over Time in Outcomes of Infants Born Less Than 30 Weeks' Gestation. Pediatrics. 2019 Sep;144(3):e20191106. doi: 10.1542/peds.2019-1106. Epub 2019 Aug 12. PMID 31405887
- [Background] Kenyon S, Boulvain M, Neilson JP. Antibiotics for preterm rupture of membranes. Cochrane Database Syst Rev. 2013 Dec 2;2013(12):CD001058. doi: 10.1002/14651858.CD001058.pub3. PMID 24297389
- [Background] Prelabor Rupture of Membranes: ACOG Practice Bulletin, Number 217. Obstet Gynecol. 2020 Mar;135(3):e80-e97. doi: 10.1097/AOG.0000000000003700. PMID 32080050
- [Background] Mercer BM, Moretti ML, Prevost RR, Sibai BM. Erythromycin therapy in preterm premature rupture of the membranes: a prospective, randomized trial of 220 patients. Am J Obstet Gynecol. 1992 Mar;166(3):794-802. doi: 10.1016/0002-9378(92)91336-9. PMID 1550145
- [Background] Mercer BM, Miodovnik M, Thurnau GR, Goldenberg RL, Das AF, Ramsey RD, Rabello YA, Meis PJ, Moawad AH, Iams JD, Van Dorsten JP, Paul RH, Bottoms SF, Merenstein G, Thom EA, Roberts JM, McNellis D. Antibiotic therapy for reduction of infant morbidity after preterm premature rupture of the membranes. A randomized controlled trial. National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. JAMA. 1997 Sep 24;278(12):989-95. PMID 9307346
- [Background] Edwards MS, Newman RB, Carter SG, Leboeuf FW, Menard MK, Rainwater KP. Randomized Clinical Trial of Azithromycin vs. Erythromycin for the Treatment of Chlamydia Cervicitis in Pregnancy. Infect Dis Obstet Gynecol. 1996;4(6):333-7. doi: 10.1155/S1064744996000671. PMID 18476121
- [Background] Hopkins S. Clinical toleration and safety of azithromycin. Am J Med. 1991 Sep 12;91(3A):40S-45S. doi: 10.1016/0002-9343(91)90401-i. PMID 1656742
- [Background] Navathe R, Schoen CN, Heidari P, Bachilova S, Ward A, Tepper J, Visintainer P, Hoffman MK, Smith S, Berghella V, Roman A. Azithromycin vs erythromycin for the management of preterm premature rupture of membranes. Am J Obstet Gynecol. 2019 Aug;221(2):144.e1-144.e8. doi: 10.1016/j.ajog.2019.03.009. Epub 2019 Mar 20. PMID 30904320
- [Background] Finneran MM, Appiagyei A, Templin M, Mertz H. Comparison of Azithromycin versus Erythromycin for Prolongation of Latency in Pregnancies Complicated by Preterm Premature Rupture of Membranes. Am J Perinatol. 2017 Sep;34(11):1102-1107. doi: 10.1055/s-0037-1603915. Epub 2017 Jun 21. No abstract available. PMID 28637060
- [Background] Pierson RC, Gordon SS, Haas DM. A retrospective comparison of antibiotic regimens for preterm premature rupture of membranes. Obstet Gynecol. 2014 Sep;124(3):515-519. doi: 10.1097/AOG.0000000000000426. PMID 25162251
- [Background] Martingano D, Singh S, Mitrofanova A. Azithromycin in the Treatment of Preterm Prelabor Rupture of Membranes Demonstrates a Lower Risk of Chorioamnionitis and Postpartum Endometritis with an Equivalent Latency Period Compared with Erythromycin Antibiotic Regimens. Infect Dis Obstet Gynecol. 2020 Jul 9;2020:2093530. doi: 10.1155/2020/2093530. eCollection 2020. PMID 32694907
- [Background] Tsai D, Jamal JA, Davis JS, Lipman J, Roberts JA. Interethnic differences in pharmacokinetics of antibacterials. Clin Pharmacokinet. 2015 Mar;54(3):243-60. doi: 10.1007/s40262-014-0209-3. PMID 25385446
- [Background] Fohner AE, Sparreboom A, Altman RB, Klein TE. PharmGKB summary: Macrolide antibiotic pathway, pharmacokinetics/pharmacodynamics. Pharmacogenet Genomics. 2017 Apr;27(4):164-167. doi: 10.1097/FPC.0000000000000270. No abstract available. PMID 28146011
- [Background] Kumar D, Moore RM, Mercer BM, Mansour JM, Redline RW, Moore JJ. The physiology of fetal membrane weakening and rupture: Insights gained from the determination of physical properties revisited. Placenta. 2016 Jun;42:59-73. doi: 10.1016/j.placenta.2016.03.015. Epub 2016 Apr 1. PMID 27238715